CLINICAL TRIAL: NCT04016493
Title: Tunnel Versus Coronally Advanced Flap Combined With a Connective Tissue Graft for the Treatment of Gingival Recessions: Long Term (4 Years) Follow-up of a Randomized Controlled Trial
Brief Title: Long-term Outcomes of Tunnel Technique
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Prof., University of Liege
Other Study IDs: H2011-1
Record Dates: First submitted 2019-06-04; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Recession, Gingival
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group (CAF+CTG; N=20)
  Interventions: Procedure: Connective tissue graft
- Test group (TUN+CTG; N=20)
  Interventions: Procedure: Connective tissue graft

INTERVENTIONS:
Procedure: Connective tissue graft — The patient received 600 mg of ibuprofen (paracetamol 1 g in case of allergy) prior to surgery, and chlorhexidine mouthwash 0.2% was provided for 2 min. Patients received local anaesthesia at the donor and recession sites (articaine hydrochloride 7200 mg/1.8 ml, adrenalin 1800 mcg/1.8 ml). CTG harvesting was performed prior to the preparation of the reception site to avoid any bias. The graft dimension was calculated according to the recession dimensions; a minimum of 3 mm of the graft was submerged mesially, distally and apically. The CTG was harvested from the palate with single edge incision and sutured with 4.0 silk. The patient was subsequently assigned randomly to the control (CAF+CTG) or the test group (TUN+CTG).

SUMMARY:
Few studies evaluate the outcomes beyond 1 year follow up for gingival recessions treatments using the tunnel technique in combination with connective tissue graft. The aim of this randomized controlled trial (RCT) was to compare the 4-year outcomes of the CAF versus the pouch/tunnel (TUN) technique both associated with CTG.

ELIGIBILITY:
Inclusion Criteria:

* Miller's class I recessions;
* Recession of 2 mm to 5 mm;
* Maxillary incisors, canines or premolars;
* Identifiable cementoenamel junction (CEJ);
* Patients minimum 18 years old;
* No/controlled periodontal disease;
* ASA1 or ASA2 (American Society of Anesthesiologists) general health status;
* Providing a signed informed consent form.

Exclusion criteria were:

* Smokers;
* Presence of cervical carious lesion;
* Pocket depth greater than 4 mm;
* Sites where previous muco-gingival therapy was performed;
* Pregnancy.
* In presence of non-carious cervical lesions, the anatomical CEJ was reconstructed by the use of a composite before the procedure.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Each patient (experimental unit) contributed a single recession. In cases of multiple recessions, the deepest one was included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Plaque Index Change | baseline, 6 months and 4 years
  The plaque accumulation is assessed at baseline, 6 months and 4 years follow-up visits using a 0-1 scoring system, 0 being the the highest value, 1 being the lowest result (0 =No detectible plaque ; 1 = Plaque can be seen by the naked eye)
Bleeding on probing score change | baseline, 6 months and 4 years
  The bleeding tendency is assessed at baseline, 6 months and 4 years follow-up visits as : 0 No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant; 1 Isolated bleeding spots visible ; 2 Blood forms a confluent red line on the margin; 3 Heavy or profuse bleeding.
Recession width change | baseline, 6 months and 4 years
  The status of the recession width was recorded at baseline, 6 months and 4 years follow-up visits.
  The scale is in mm. More large is it, worst it is Minest large it is, best it is
Gingival thickness change | baseline, 6 months and 4 years
  The gingival thickness was recorded at baseline, 6 months and 4 years follow-up visits.
  The scale is in mm. More thick is it, best it is Minest thick it is, worst it is
Keratinised mucosa height change | baseline, 6 months and 4 years
  The status of the keratinised mucosa height was recorded at baseline, 6 months and 4 years follow-up visits.
  The scale is in mm. More large is it, best it is Minest large it is, worst it is
Mean Root Coverage change | at 6 months and 4 years.
  The status of the Mean Root Coverage was recorded at 6 months and 4 years follow-up visits.
  The scale is in mm. More long it is, best it is Minest long it is, worst it is
PES Assessment change | Baseline, 6 months and 4 years
  The PES was assessed according to the seven parameters described by Fürhauser (Fürhauser et al., 2005).

SECONDARY OUTCOMES:
Patient-related esthetic outcomes | 4 years
  (Fürhauser et al., 2005). Patient-related esthetic outcomes were also recorded in a questionnaire using a 0-14 graduated scale (0 being the worst and 14 the best value).

IPD SHARING:
Plan to Share IPD: Undecided